CLINICAL TRIAL: NCT02635477
Title: Get Going: Fellow-Led Trial of an Accelerometer-Based Intervention to Promote Physical Activity in Frail Older Adults Transitioning From a Cardiovascular Hospitalization to Home
Brief Title: Get Going: Accelerometer-Based Intervention to Promote Physical Activity in Frail Older Adults
Acronym: AAIMASP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American College of Cardiology (Other)
Collaborators: Alliance for Academic Internal Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAIM ASP 2015
Record Dates: First submitted 2015-10-28; First posted 2015-12-18 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2016-11

CONDITIONS: Coronary Artery Disease; Heart Failure
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): frail elderly patients discharged from a cardiovascular hospitalization; provided with an actigraphy device that displays an adaptive personalized daily step count goal and audible alerts to increase physical activity
  Interventions: Behavioral: Intervention
- Control Group (Experimental): frail elderly patients discharged from a cardiovascular hospitalization; provided with a matching actigraphy device that has a blacked-out screen and does not display step count goals or provide audible alerts (functions in silent monitoring mode only)
  Interventions: Behavioral: Intervention; Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — Behavioral: actigraphy device, adaptive step count algorithm
Behavioral: Control — Behavioral: actigraphy device, step count measurement only
  Arms: Control Group

SUMMARY:
A multicenter prospective randomized clinical trial testing the hypothesis that a patient-centered actigraphy intervention will result in increased physical activity for frail older adults increase during the critical first 30 days after a cardiovascular hospitalization.

DETAILED DESCRIPTION:
The transition from hospital to home is critical for older patients after a cardiovascular hospitalization, since 1 in 3 will suffer the fate of functional decline or repeat hospitalizations within the first 30 days. This has a tremendous impact on the patient, leading to a vicious cycle of worsening health status and disability, and the healthcare system, leading to an estimated $12 billion of preventable costs. At the policy level, preventing readmissions has become a national priority at the forefront of the medical agenda.

Frailty, a geriatric syndrome characterized by subclinical impairments in multiple organs and decreased physiologic resiliency, is a major risk factor for unsuccessful transitions of care and adverse health outcomes. Thus, it has been suggested that interventions aimed at improving transitions of care should target frail patients. Frail individuals demonstrate a well-defined phenotype of muscle weakness and physical inactivity, readily measurable using various scales and instruments. To date, the most widely studied intervention to improve frailty and related outcomes has been physical activity.

However, fewer than 50% of patients adhere to regular physical activity programs. Enrollment in cardiac rehabilitation programs is even lower owing to multiple barriers, including lack of payer reimbursement ≤ 30 days after a hospitalization, the highest risk period for readmissions. Scientific statements have called for augmented "self-care" to assure adequate physical activity in patients with heart failure and other forms of cardiovascular disease 10. Moreover, low-intensity home-based physical activity programs can be as efficacious as higher-intensity center-based programs, strengthening the rationale for self-care.

The advent of small, portable, inexpensive accelerometer devices has emerged as a powerful tool to facilitate self-monitored physical activity. These devices are worn by patients and provide real-time feedback about the number of steps walked each day (as well as other functional parameters). This is in tune with a systematic review which found that feedback and goal setting improved adherence to physical activity in patients with heart failure. A few studies in the physical therapist literature have used accelerometers to demonstrate low baseline physical activity and boost total step counts in patients attending cardiac rehabilitation, but these patients were at least 30 days removed from their index hospitalization, and none enrolled patients in the critical post-discharge phase.

Research question: Is a portable actigraphy-based intervention more effective than standard-of-care in promoting physical activity in the first 30 days after hospital discharge among frail older adults with cardiovascular disease?

ELIGIBILITY:
Inclusion Criteria:

1. older adults aged ≥70 years,
2. at least one criteria positive on the FRAIL scale,
3. hospital discharge to an independent residence,
4. primary final discharge diagnosis of coronary disease or heart failure but not requiring cardiac surgery or TAVR during the index hospitalization,
5. able to stand and walk without assistance from another person,
6. able to carry out basic activities of daily living without assistance as per Clinical Frailty Scale rating ≤5,
7. signed informed consent from the patients, and
8. approval from the treating physician that the patient is safe and appropriate to participate in this trial.

Exclusion Criteria:

1. cognitive impairment defined by a positive mini-cog test or known moderate or severe dementia,
2. more than one fall in the past six months, or a fall in the past three months prior to hospitalization,
3. high-risk for falls or unsteady for mobilization according to a clinical physical therapist's assessment (if performed) or as assessed during functional testing,
4. non-revascularized acute myocardial infarction within the past month (unless revascularization was not indicated) or uncorrected severe symptomatic aortic stenosis,
5. active severe symptoms of angina, dyspnea, or claudication at rest or with minimal activity (Canadian Cardiovascular Society class 4, New York Heart Association class 4, or Fontaine class 3-4, respectively),
6. referral to a structured cardiac rehabilitation program in the first 30 days after hospital discharge (not counting home-based physical therapy),
7. unable to return for follow-up visit, and
8. poor comprehension of the actigraphy device.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Steps taken per day | 1 year
  The primary outcome measure for this study is the average number of steps walked per day during the study period (excluding the run-in phase), as determined by the actigraphy device.

SECONDARY OUTCOMES:
Quality of life | baseline, 30 days
  A secondary outcome for this study is quality of life, as determined by score on the EQ-5D questionnaire
Short physical performance battery | baseline, 30 days
  A secondary outcome for this study is physical performance, as determined by the change in Short Physical Performance Battery score from baseline to 30-days.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hummel, MD, Principal Investigator — University of Michigan Ann Arbor, Michigan, USA; Jonathan Afilalo, MD, MSc, Principal Investigator — Jewish General Hospital, McGill University, Montreal, Quebec, Canada
Locations (16):
- United States (14):
  - Emory University, Atlanta, Georgia
  - Boston Veterans Affairs, Boston, Massachusetts
  - Ann Arbor Veterans Affairs, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - Beaumont Health System/Oakwood, Dearborn, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - Mayo Clinic, Rochester, New Hampshire
  - New York Presbyterian Hospital/Columbia, New York, New York
  - New York Presbyterian Hospital/Cornell, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University/University Hospital, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington
- Canada (2):
  - McGill University, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec

REFERENCES:
- [Result] Goldwater DS. Geriatric cardiology: a fellow's perspective. J Am Coll Cardiol. 2014 Sep 30;64(13):1401-3. doi: 10.1016/j.jacc.2014.08.009. No abstract available. PMID 25257643
- [Result] Martin SS, Ou FS, Newby LK, Sutton V, Adams P, Felker GM, Wang TY. Patient- and trial-specific barriers to participation in cardiovascular randomized clinical trials. J Am Coll Cardiol. 2013 Feb 19;61(7):762-9. doi: 10.1016/j.jacc.2012.10.046. PMID 23410547
- [Result] Gurwitz JH. The exclusion of older people from participation in cardiovascular trials. Virtual Mentor. 2014 May 1;16(5):365-8. doi: 10.1001/virtualmentor.2014.16.05.pfor1-1405. No abstract available. PMID 24847706
- [Result] Afilalo J, Eisenberg MJ, Morin JF, Bergman H, Monette J, Noiseux N, Perrault LP, Alexander KP, Langlois Y, Dendukuri N, Chamoun P, Kasparian G, Robichaud S, Gharacholou SM, Boivin JF. Gait speed as an incremental predictor of mortality and major morbidity in elderly patients undergoing cardiac surgery. J Am Coll Cardiol. 2010 Nov 9;56(20):1668-76. doi: 10.1016/j.jacc.2010.06.039. PMID 21050978
- [Result] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966
- [Result] Lindman BR, Alexander KP, O'Gara PT, Afilalo J. Futility, benefit, and transcatheter aortic valve replacement. JACC Cardiovasc Interv. 2014 Jul;7(7):707-16. doi: 10.1016/j.jcin.2014.01.167. Epub 2014 Jun 18. PMID 24954571
- [Result] Afilalo J, Alexander KP, Mack MJ, Maurer MS, Green P, Allen LA, Popma JJ, Ferrucci L, Forman DE. Frailty assessment in the cardiovascular care of older adults. J Am Coll Cardiol. 2014 Mar 4;63(8):747-62. doi: 10.1016/j.jacc.2013.09.070. Epub 2013 Nov 27. PMID 24291279
- [Result] Forman DE, Rich MW, Alexander KP, Zieman S, Maurer MS, Najjar SS, Cleveland JC Jr, Krumholz HM, Wenger NK. Cardiac care for older adults. Time for a new paradigm. J Am Coll Cardiol. 2011 May 3;57(18):1801-10. doi: 10.1016/j.jacc.2011.02.014. No abstract available. PMID 21527153
- [Result] Riegel B, Moser DK, Anker SD, Appel LJ, Dunbar SB, Grady KL, Gurvitz MZ, Havranek EP, Lee CS, Lindenfeld J, Peterson PN, Pressler SJ, Schocken DD, Whellan DJ; American Heart Association Council on Cardiovascular Nursing; American Heart Association Council on Cardiovascular Nursing; American Heart Association Council on Clinical Cardiology; American Heart Association Council on Nutrition, Physical Activity, and Metabolism; American Heart Association Interdisciplinary Council on Quality of Care and Outcomes Research. State of the science: promoting self-care in persons with heart failure: a scientific statement from the American Heart Association. Circulation. 2009 Sep 22;120(12):1141-63. doi: 10.1161/CIRCULATIONAHA.109.192628. Epub 2009 Aug 31. No abstract available. PMID 19720935
- [Result] King AC, Haskell WL, Taylor CB, Kraemer HC, DeBusk RF. Group- vs home-based exercise training in healthy older men and women. A community-based clinical trial. JAMA. 1991 Sep 18;266(11):1535-42. PMID 1880885
- [Result] Hwang R, Marwick T. Efficacy of home-based exercise programmes for people with chronic heart failure: a meta-analysis. Eur J Cardiovasc Prev Rehabil. 2009 Oct;16(5):527-35. doi: 10.1097/HJR.0b013e32832e097f. PMID 20054288
- [Result] Tierney S, Mamas M, Woods S, Rutter MK, Gibson M, Neyses L, Deaton C. What strategies are effective for exercise adherence in heart failure? A systematic review of controlled studies. Heart Fail Rev. 2012 Jan;17(1):107-15. doi: 10.1007/s10741-011-9252-4. PMID 21567221
- [Result] Savage PD, Ades PA. Pedometer step counts predict cardiac risk factors at entry to cardiac rehabilitation. J Cardiopulm Rehabil Prev. 2008 Nov-Dec;28(6):370-7; quiz 378-9. doi: 10.1097/HCR.0b013e31818c3b6d. PMID 19008690
- [Result] Izawa KP, Watanabe S, Hiraki K, Morio Y, Kasahara Y, Takeichi N, Oka K, Osada N, Omiya K. Determination of the effectiveness of accelerometer use in the promotion of physical activity in cardiac patients: a randomized controlled trial. Arch Phys Med Rehabil. 2012 Nov;93(11):1896-902. doi: 10.1016/j.apmr.2012.06.015. Epub 2012 Jun 28. PMID 22750166
- [Result] Bravata DM, Smith-Spangler C, Sundaram V, Gienger AL, Lin N, Lewis R, Stave CD, Olkin I, Sirard JR. Using pedometers to increase physical activity and improve health: a systematic review. JAMA. 2007 Nov 21;298(19):2296-304. doi: 10.1001/jama.298.19.2296. PMID 18029834
- [Result] Vaes AW, Cheung A, Atakhorrami M, Groenen MT, Amft O, Franssen FM, Wouters EF, Spruit MA. Effect of 'activity monitor-based' counseling on physical activity and health-related outcomes in patients with chronic diseases: A systematic review and meta-analysis. Ann Med. 2013 Sep;45(5-6):397-412. doi: 10.3109/07853890.2013.810891. Epub 2013 Jul 3. PMID 23952917
- [Result] Izawa KP, Watanabe S, Oka K, Hiraki K, Morio Y, Kasahara Y, Brubaker PH, Osada N, Omiya K, Shimizu H. Usefulness of step counts to predict mortality in Japanese patients with heart failure. Am J Cardiol. 2013 Jun 15;111(12):1767-71. doi: 10.1016/j.amjcard.2013.02.034. Epub 2013 Mar 27. PMID 23540653
- [Result] Cyarto EV, Myers A, Tudor-Locke C. Pedometer accuracy in nursing home and community-dwelling older adults. Med Sci Sports Exerc. 2004 Feb;36(2):205-9. doi: 10.1249/01.MSS.0000113476.62469.98. PMID 14767241
- [Result] Nguyen HQ, Steele BG, Dougherty CM, Burr RL. Physical activity patterns of patients with cardiopulmonary illnesses. Arch Phys Med Rehabil. 2012 Dec;93(12):2360-6. doi: 10.1016/j.apmr.2012.06.022. Epub 2012 Jul 5. PMID 22772084
- [Result] Leidy NK, Kimel M, Ajagbe L, Kim K, Hamilton A, Becker K. Designing trials of behavioral interventions to increase physical activity in patients with COPD: insights from the chronic disease literature. Respir Med. 2014 Mar;108(3):472-81. doi: 10.1016/j.rmed.2013.11.011. Epub 2013 Nov 20. PMID 24315467